CLINICAL TRIAL: NCT04523441
Title: Identification of the Needs and Difficulties Associated With the Perceptual-motor Management of Infants at High Risk of Cerebral Palsy During the First 24 Months Following Neonatal Hospitalization. Qualitative Study Among Parents and Health Professionals
Brief Title: Early Support and Physiotherapy for Children and Their Motor Skills
Acronym: App-eMot-Quali
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: KRUMM APPARA 2019
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Infant; Cerebral Palsy; Neonatal
MeSH Terms: conditions — Cerebral Palsy | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents: man or woman
  Interventions: Other: Semi-directive interview
- Professionals: health professionals in charge of monitoring children
  Interventions: Other: Focus group

INTERVENTIONS:
Other: Focus group — Holding of a focus group by a sociologist
  Groups: Professionals
Other: Semi-directive interview — Conducting a semi-directive interview by a sociologist after discharge from hospital
  Groups: Parents

SUMMARY:
The App-eMot-Quali project proposed here is the first phase in the implementation of a care pathway supported by a digital tool. It consists of a qualitative study allowing individual interviews to be conducted with parents of infants at high risk of cerebral palsy and health professionals in order to identify and precisely describe the needs and difficulties present during the child's rehabilitative care during the first months of life.

ELIGIBILITY:
Inclusion Criteria:

1. For the parents:

   Parents of children under 24 months of age at high risk of cerebral palsy who have given their oral consent.

   Children at high risk of cerebral palsy are defined as :
   * Premature children ≤ 31 WG + 6 days or birth weight less than 1000g.
   * Children who have had a stroke or stage 2 or 3 hypoxia-ischemia according to the Sarnat classification.

   The selection of parents may be retrospective with less than 24 months since hospital discharge.
2. For the health professionals:

Physiotherapists, psychomotricians, psychologists and doctors involved in the care of children at high risk of cerebral palsy.

Exclusion Criteria:

* A person who is physically or cognitively unable to participate in a one-on-one interview or who does not have a sufficient command of the French language.
* Parents aged <18 years
* Parents in protective custody
* Parents of children with major orthopedic or traumatic disorders unrelated to the high risk of cerebral palsy.
* Parents of a child with a genetic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents of children under 24 months of age and health professionals working in the paediatric intensive care unit at the Dijon Bougogne University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Typology and categorization of the needs and difficulties encountered by the parents. | Through study completion an average of 21 months
  collected through semi-directive individual interviews with parents

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France